CLINICAL TRIAL: NCT06679088
Title: GlyCoBrain Observation - Breakfast Habits Among Students With Early and Late Chronotype
Brief Title: GlyCoBrain Observational Study
Acronym: GlyCoBrainOb
Status: Enrolling by invitation | Type: Observational
Sponsor: Paderborn University (Other)
Responsible Party: Principal Investigator, Anette Buyken, Prof. Dr. Anette Buyken, Head of the research group "Public Health Nutrition", Paderborn University
Other Study IDs: BU 1807/8-1
Record Dates: First submitted 2024-11-05; First posted 2024-11-07 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2024-11

CONDITIONS: Healthy; Adult
Keywords: Chronotype; Breakfast; Glyceamic Index; MCTQ; Academic performance; Dietary patterns; Student nutrition; Nutrient composition

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- students of Paderborn University: 18 years to 25 years (adult)

SUMMARY:
Breakfasts with a high glycaemic index (GI) resulting in sharp rises in blood glucose may adversely affect memory and attention, particularly in the late postprandial phase (i.e., 120-180 minutes after breakfast). Young adults may be particularly responsive to these adverse effects on cognition since they are prone to experience circadian misalignment because their midpoint of sleep (i.e., chronotype) is biologically most delayed in young adulthood. Our recent research suggests that persons with a later chronotype exhibit no diurnal difference in response to a high GI meal consumed in the morning and evening, suggesting that consumption of an early breakfast "against the inner clock" may be adverse for their glycaemic response and that consumption of an early breakfast may present a burden for those with a later chronotype. Indeed, persons with later chronotypes commonly tend to exhibit less favourable eating pattern. Hence, consuming an early breakfast, e.g. in preparation for an exam, may be more problematic for persons with later chronotypes and it may be more likely that these persons choose less favorable foods for breakfast.

Thus, it remains to be clarified whether persons with a later chronotype:

1. usually consume breakfasts with a higher dietary GI than those with an earlier chronotype. Addressing this hypothesis needs to consider both the first and second breakfast (i.e., all meals until noon), since breakfast skipping may be common particularly among persons with a later chronotype
2. are more prone to consume foods from higher GI sources in preparation for an exam in the morning than those with an earlier chronotype.
3. consume breakfasts of a higher energy density and a lower micronutrient adequacy than persons with an earlier chronotype.

In this study (GlyCoBrain (Glycaemic index Cognition Brain) observational study), 350 students from the University of Paderborn, aged between 18 and 25, will be recruited until the end of February 2025. A questionnaire-based screening will assess breakfast habits and chronotype using the Munich ChronoType Questionnaire (MCTQ). In addition, students will be asked to fill in two 24-h recalls (myFood24) to provide information on their habitual diet (including breakfast). The screening will be followed by two controlled intervention studies examining the effect of (i) a high GI breakfast (GlyCoBrain intervention study 1) and (ii) a breakfast causing an (isolated) reactive hypoglycaemia (GlyCoBrain intervention study 2) on the course of memory and attention in the postprandial phase.

DETAILED DESCRIPTION:
Background Breakfast is commonly considered one of the most important meals of the days. Failure to consume a breakfast, i.e., breakfast skipping, has been related to an increased risk of overweight/obesity or type 2 diabetes in the longer-term, but may also adversely affect cognition and academic performance. Similarly, breakfasts with a high glycaemic index (GI) resulting in sharp rises in blood glucose may adversely affect memory and attention, particularly in the late postprandial phase (i.e., 120-180 minutes after breakfast). A recent meta-analysis suggests specific effects for immediate and delayed episodic memory among persons with a better glucose tolerance.

Whilst young adults generally have a better glucose tolerance they are, however, prone to circadian misalignment since their midpoint of sleep (i.e., chronotype) is most delayed. Chronotype is a biological construct mainly influenced by genetics, sex and age. Chronotype tends to shift later from adolescence into early adulthood with the peak of delay around age 20 before moving back to an earlier chronotype. Hence, persons in young adulthood are more likely to have a later chronotype and experience a circadian misalignment between the "inner clock" and social requirements. Such a desynchronization may lead to poorer glucose tolerance and an exaggerated glucose response to a high GI breakfast in individuals with a later chronotype. Our recent research suggests that persons with a later chronotype were similarly vulnerable to both very early and late high GI meals, whereas earlier chronotypes had lower glucose responses to the high GI meal consumed at breakfast. In addition, research from female twins suggests that timing of breakfast has a larger underlying genetic component than timing of dinner, suggesting that consumption of an early breakfast may present a burden for those with a later chronotype. As a result, the cognitive performance of people with a later chronotype could particularly benefit from consuming a low GI breakfast. Current studies also report that later chronotypes delay their meal timing, tend to skip breakfast, are at higher risk to consume larger meals at night than earlier chronotypes and to have less favourable dietary pattern, consuming less protein and vegetables and more sweets, sugar, alcohol and coffee.

Taken together, a later chronotype may make young adults more vulnerable to consume unfavourable breakfasts, i.e. breakfasts with a higher dietary GI, higher energy density and lower micronutrient adequacy. However, to date no study has investigated breakfast habits in relation to chronotype in young adults. Furthermore, it remains to be elucidated which food students choose to account for the necessity of academic performance in preparation for an exam in the morning.

The present study will examine the relevance of breakfast among students in detail and relate this to their chronotype. The observational study will be followed by two nutritional intervention studies only with the earliest and latest chronotypes to examine the effects of high GI breakfast or a breakfast causing a reactive hypoglycaemia on cognitive functions in the early morning.

Hypothesis The hypothesis of the GlyCoBrain observational study is that students with a later chronotype are more likely to consume breakfasts with a higher dietary GI, higher breakfast energy density and lower breakfast micronutrient adequacy. We also postulate that persons with a later chronotype are more prone to consume foods from higher GI sources in preparation for an exam than those with an earlier chronotype.

Aim The aim of the GlyCoBrain observational study is to investigate the breakfast habits of German students aged 18-25 years in relation to their chronotype.

Methods 1 (Participants): The researchers will initially recruit at least 350 students aged 18 to 25 from the University Paderborn who meet the specified inclusion criteria (see Participation Criteria). Recruitment and screening are planned to take place from October 2024 until the end of February 2025. Using the GlyCoBrain observational study, participants with the earliest and latest chronotypes will be identified for subsequent inclusion in the GlyCoBrain intervention studies.

Methods 2 (Methods): In the screening of the GlyCoBrain observational study, participants are first asked to provide general information (gender, age, university schedule, time of last menstruation). Additionally, the criteria for exclusion from participation in the screening of the observational study as well as the intervention studies are queried. This includes information on smoking status, shift work, travel across more than two time zones in the past three months, pregnancy, breastfeeding, medication use, chronic diseases, food intolerances, and allergies. Chronotype, that is defined as the midpoint of the sleep period (mid-time sleep), will be assessed with the Munich ChronoType questionnaire (MCTQ, © Roenneberg and co-workers, 2015). To assess the Chronotype, participants will be asked about their sleep behavior over the past four weeks. Sleep patterns on workdays and free days are inquired about separately to account for differences in sleep duration and timing. This separation is important for accurately adjusting the chronotype calculation, considering differences in sleep duration and timing between these days. In the MCTQ, students will be asked whether they engage in regular work (including study periods), how many days they perform this activity, when they go to bed, how long it takes them to fall asleep, when they wake up, and when they get up.

In addition, the breakfast behavior on exam days will be surveyed in comparison to normal days on which lectures will take place. The questionnaire assumes that the exam is taken at 9 o'clock to simulate a realistic daily routine. The breakfast behavior questionnaire evaluates the extent to which a participants' intake of specific food (29 items), beverages (14 items), meal replacements, or supplements on exam days differs from that on regular days. Participants are also asked where and at what time they eat their breakfast. Further, students will be asked to provide information about any food allergies and details on the food and beverages they bring to the exam.

Habitual intake is assessed by two 24-hour recalls, one collected at the study center at the day of the visit and another one collected remotely at home within 1 week from the visit. The German version of myFood24, a web-based dietary assessment tool, will be used for accurately capturing individuals' dietary intake. In myFood24, students are required to input detailed information about the foods and beverages they have consumed on the day before, including portion sizes and meal types. This data is then analyzed against a food composition database to provide insights into nutrient intake and dietary patterns.

Additionally, body composition will be assessed by Bioimpedance Analysis (BIA, mBCA 515, SECA) to estimate individual percentages of body fat, muscle mass, total body water and extracellular water. Additionally, body weight is measured directly by the medical Body Composition Analyzer (mBCA). Body height is measured using an ultrasound measuring station (seca 287 db). Waist circumference is assessed on the exposed upper body at the midpoint between the lower ribcage and the hip bone. Furthermore, information on physical activity (using a questionnaire from the Study on "Health in Adults in Germany", part of the Robert-Koch-Institut (RKI, Germany)) and screen-time (using a questionnaire previously employed in the Dortmund Nutritional and Anthropometric Longitudinally Designed (DONALD) study, a long-term observational study at University Bonn, Germany) will be collected.

Statistical analyses Multivariable multilevel regression models will be used to examine whether a later chronotype is associated with a less favorable breakfast GI, breakfast food choices and breakfast energy density and nutrient composition. Models will adjust for potential confounders (e.g., sex, age, life-style characteristics, body composition).

ELIGIBILITY:
Inclusion Criteria:

* Students at Paderborn University aged between 18 and 25 years
* Proficient in the German language because all questionnaires are in German.

Exclusion Criteria:

* Students studying nutritional science and home economics
* acute or permanent use of sleep-promoting medications (including herbal preparation):
* chemical medications: melatonin, diphenhydramine, doxylamine
* herbal preparations: hops, St. John's wort, lemon balm, lavender, passionflower, Baldurat, Neurexan, cannabinoids
* Use of psychotropic medications (antidepressants, tranquilizer, antipsychotics)
* Use of methylphenidate (e.g. Ritalin, Medikinet, Concerta)
* Use of cannabinoids by prescription
* Continuous administration of antihistamines when discontinuation is not feasible during the intervention
* Use of herbal preparations affecting memory and concentration (e.g. gingko, ginseng, ashwagandha)
* Use of other medications (e.g. insulin, metformin, SGLT2 inhibitors, steroids, ACE inhibitors)
* Selected chronic diseases (depression and other mental disorders such as anxiety disorder, ADHD, diabetes mellitus (all types), prediabetes, blood clotting disorders (e.g., thrombocytopenia, hemophilia), eating disorders (e.g., anorexia, binge eating, bulimia)
* Addiction disorders (e.g., alcohol, drug, or medication dependency)
* Chronic inflammatory bowel diseases
* infectious diseases (HIV, hepatitis)
* Pregnant and breastfeeding individuals
* Shift work or travel in the past 3 months across more than 2 time zones
* students with a pacemaker/defibrillator

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Students at Paderborn University (see inclusion criteria)
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Breakfast quality, dietary GI and nutrient composition | At inclusion into the study and after 6 days
  2 times Computer-assisted 24-hour recall of consumed foods and beverages in the past 24 h
Breakfast food choice in preparation of an exam | Assessed once at the beginning of the study
  Questionnaire inquiring selected food items, beverages and meal replacements

CONTACTS AND LOCATIONS:
Locations (1):
- Paderborn University, Paderborn, North-Rhine-Westfalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Koch SAJ, Conrad J, Cade JE, Weinhold L, Alexy U, Nothlings U. Validation of the web-based self-administered 24-h dietary recall myfood24-Germany: comparison with a weighed dietary record and biomarkers. Eur J Nutr. 2021 Oct;60(7):4069-4082. doi: 10.1007/s00394-021-02547-7. Epub 2021 May 11. PMID 33974128
- [Background] Koch SAJ, Conrad J, Hierath L, Hancock N, Beer S, Cade JE, Nothlings U. Adaptation and Evaluation of Myfood24-Germany: A Web-Based Self-Administered 24-h Dietary Recall for the German Adult Population. Nutrients. 2020 Jan 6;12(1):160. doi: 10.3390/nu12010160. PMID 31935885
- [Background] Nowack K, Van Der Meer E. The synchrony effect revisited: chronotype, time of day and cognitive performance in a semantic analogy task. Chronobiol Int. 2018 Nov;35(12):1647-1662. doi: 10.1080/07420528.2018.1500477. Epub 2018 Aug 7. PMID 30085831
- [Background] Xiao Q, Garaulet M, Scheer FAJL. Meal timing and obesity: interactions with macronutrient intake and chronotype. Int J Obes (Lond). 2019 Sep;43(9):1701-1711. doi: 10.1038/s41366-018-0284-x. Epub 2019 Jan 31. PMID 30705391
- [Background] Pengpid S, Peltzer K. Skipping Breakfast and Its Association with Health Risk Behaviour and Mental Health Among University Students in 28 Countries. Diabetes Metab Syndr Obes. 2020 Aug 18;13:2889-2897. doi: 10.2147/DMSO.S241670. eCollection 2020. PMID 32884315
- [Background] Ballon A, Neuenschwander M, Schlesinger S. Breakfast Skipping Is Associated with Increased Risk of Type 2 Diabetes among Adults: A Systematic Review and Meta-Analysis of Prospective Cohort Studies. J Nutr. 2019 Jan 1;149(1):106-113. doi: 10.1093/jn/nxy194. PMID 30418612
- [Background] Ma X, Chen Q, Pu Y, Guo M, Jiang Z, Huang W, Long Y, Xu Y. Skipping breakfast is associated with overweight and obesity: A systematic review and meta-analysis. Obes Res Clin Pract. 2020 Jan-Feb;14(1):1-8. doi: 10.1016/j.orcp.2019.12.002. Epub 2020 Jan 7. PMID 31918985
- [Background] Gibney MJ, Barr SI, Bellisle F, Drewnowski A, Fagt S, Livingstone B, Masset G, Varela Moreiras G, Moreno LA, Smith J, Vieux F, Thielecke F, Hopkins S. Breakfast in Human Nutrition: The International Breakfast Research Initiative. Nutrients. 2018 May 1;10(5):559. doi: 10.3390/nu10050559. PMID 29723985
- [Background] Kanerva N, Kronholm E, Partonen T, Ovaskainen ML, Kaartinen NE, Konttinen H, Broms U, Mannisto S. Tendency toward eveningness is associated with unhealthy dietary habits. Chronobiol Int. 2012 Aug;29(7):920-7. doi: 10.3109/07420528.2012.699128. PMID 22823875
- [Background] Mazri FH, Manaf ZA, Shahar S, Mat Ludin AF. The Association between Chronotype and Dietary Pattern among Adults: A Scoping Review. Int J Environ Res Public Health. 2019 Dec 20;17(1):68. doi: 10.3390/ijerph17010068. PMID 31861810
- [Background] Stutz B, Krueger B, Goletzke J, Jankovic N, Alexy U, Herder C, Dierkes J, Berg-Beckhoff G, Jakobsmeyer R, Reinsberger C, Buyken AE. Glycemic response to meals with a high glycemic index differs between morning and evening: a randomized cross-over controlled trial among students with early or late chronotype. Eur J Nutr. 2024 Aug;63(5):1593-1604. doi: 10.1007/s00394-024-03372-4. Epub 2024 Apr 12. PMID 38605233
- See also: The main aspects of the observational study are described on the website. Information is provided on the aim of the study, eligibility criteria and information on the subsequent intervention study with the data to be collected. — https://sug.uni-paderborn.de/ekg/glycobrain